CLINICAL TRIAL: NCT04172480
Title: HUSH Restriction in HIV Infected Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS RF 004
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC conserved in RLT Buffer for viral DNA and RNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- acute HIV1 infection: Patient infected by HIV1, prior treatment initiation
  Interventions: Other: Blood sampling
- chronic HIV1 infection: Patient infected by HIV1, untreated or without treatment since at least 3 months
  Interventions: Other: Blood sampling
- HIV2 infection: Patient infected by HIV2, untreated or without treatment since at least 3 months
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Peripheral blood sampling on EDTA

SUMMARY:
HIV eradication faces a major obstacle that is viral persistence in latent reservoir cells despite antiretroviral therapy. Epigenetic repression plays a central role in viral transgene latency and several epigenetic regulators have been involved in this process. Among them, the "Human Silencing Hub" or HUSH complex, composed of Tasor, MPP8 and periphilin, has been shown to recruit the H3K9me3 methyltransferase "SET domain bifurcated 1" (SETDB1) and is therefore responsible for genes' epigenetic repression. Our recent results highlight the ability of Vpx from HIV-2/SIVsmm to counteract HUSH and to reactivate latent viruses in a latency model. We propose here to study HUSH activity along pathogenesis.

ELIGIBILITY:
Inclusion Criteria for group 1:

* Symptomatic or asymptomatic acute HIV1 infection
* Age above 15 years old
* No ARV treatment prior inclusion (excepted as prophylaxis pre or post exposure)

Inclusion Criteria for group 2:

* Chronic HIV1 infection
* Age above 18 years old
* No ARV treatment since at least 3 month (regardless the reason)

Inclusion Criteria for group 3:

* HIV2 Infection
* Age above 18 years old
* No ARV treatment since at least 3 month (regardless the reason)

Exclusion Criteria for all groups:

* HIV1 and HIV2 co-infection
* Evolutive intercurrent pathology, in particular active co-infection (i.e. HBV, HCV, tuberculosis, HTLV1)
* Life-threatening pathology

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population infected either by HIV1 or HIV2
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Viremia | Baseline
  Intracellular HIV RNA load expressed in number of copies / ml
Total HIV DNA and integrated HIV DNA | Baseline
  Quantification by qPCR
Hush activity | Baseline
  Transcription rate of cellular genes targeted by HUSH by qRT-PCR

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôtel-Dieu, Paris
  - Hôpital Necker, Paris